CLINICAL TRIAL: NCT02983682
Title: A Pilot Study of the Effectiveness of Lidocaine Infusions for the Management of Chronic Pain in Children
Brief Title: Lidocaine Infusions for Chronic Pain in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lisa Isaac, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000052256
Record Dates: First submitted 2016-04-15; First posted 2016-12-06 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pain, Chronic
Keywords: Anesthetics, Local; Lidocaine; Pediatrics; Children; Adolescents
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lidocaine Infusion (Experimental): All participants will receive intravenous lidocaine infusion of 42 mcg/kg/minute over 2 hours, for a total of 5 mg/kg. No bolus dose will be given.
  Interventions: Drug: Lidocaine Infusion

INTERVENTIONS:
Drug: Lidocaine Infusion — Patients will receive lidocaine infusion of 42 micrograms/kg/minute over tow hours for a total of 5 mg/kg.
  Other Names: Preservative Free Lidocaine Hydrochloride

SUMMARY:
This is a study to evaluate the efficacy and safety of lidocaine in the management of chronic pain in children. All participants will receive lidocaine infusion and severity of pain and degree of chronic-pain related disability will be assessed before and up to 4 weeks after infusion. Adverse events will be recorded.

DETAILED DESCRIPTION:
Reports have shown that intravenous lidocaine infusions have been effective in relieving chronic pain that has been resistant to other therapies, with minimal side effects. The investigators would like to determine whether severity of pain and degree of chronic-pain related disability could be reduced with lidocaine infusion in children and to understand whether the dose of lidocaine correlates with blood levels in the same manner as it does in adults. The investigators will recruit 24 patients aged 8-18 with chronic pain that has not been relieved by standard therapies. Each patient will receive a lidocaine infusion over 2 hours. Blood will be drawn for lidocaine concentration before the beginning of the infusion, immediately after and 0.5, 2 and 4 hours after. Severity of pain and degree of disability will be recorded using a questionnaire measuring pain scores, sleep disruption, social disruption, physical abilities and school attendance before the infusion, weekly for 2 weeks and then 4 weeks after. This study will help the investigators better understand the effectiveness and safety of intravenous lidocaine for chronic pain in children.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a chronic pain condition (> 3 months) other conventional medical therapies (anticonvulsants, tricyclics etc), have not been effective.
2. American Society of Anesthesiologists class 1 or 2
3. Age 8-18 years
4. Ability to understand and use the numeric rating scale to rate their pain and to understand and answer other questionnaires
5. Negative pregnancy test in participants of child-bearing potential (Females 12 years of age and older, or menarchal if under 12)

Exclusion Criteria:

1. History of seizures
2. Known liver or renal disease
3. Patient taking strong CYP1A2 inducers or inhibitors (fluvoxamine, phenytoin, cimetidine, amiodarone) or beta blockers (propranolol, metoprolol, nadolol)
4. Allergy or sensitivity to lidocaine or other local anesthetic
5. Cardiac conduction anomalies (eg. Heart block, Wolff-Parkinson-White)
6. Serum electrolytes (potassium, sodium, magnesium or calcium) outside of reference ranges
7. Pregnancy

Withdrawal Criteria

1. Patient or parent/guardian request
2. Refusal to have intravenous access and serum levels drawn
3. Inability to complete pain scores on the questionnaires (paper or electronic) at the first infusion and weekly for 2 weeks and at one month following infusion
4. Baseline free carnitine concentration < 26 micromoles/L or total carnitine < 32 micromoles/L (reference values from SickKids Department of Pediatric Laboratory Medicine "Guide to Laboratory Services")

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Pain Score | Change from baseline pain score (7 days prior to infusion) at 14 days after completion of infusion
  Pain scores will be measured using the Numeric Rating Scale

SECONDARY OUTCOMES:
Analgesic Requirement | Up to seven days prior to lidocaine infusion.
  Participants will record all analgesics used in a pain diary provided by the investigators.
Analgesic Requirement | Up to one month after lidocaine infusion
  Participants will record all analgesics used in a pain diary provided by the investigators.
Adverse Events | intraoperative
  Participants will be monitored for adverse events including cardiac arrhythmias, hypotension, hypertension, tachycardia, metallic taste, tinnitus, lightheadedness, nausea, vomiting and headache

OTHER OUTCOMES:
Sleep | Day of the infusion, one week, two weeks and four weeks following the infusion.
  The Adolescent Sleep Wake Scale will be used to assess quantity and quality of sleep.
Pain Interference | Day of the infusion, one week, two weeks and four weeks following infusion.
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale will be used to measure how pain interferes with the participants activities of daily living
School Attendance | Week prior to the infusion and at two and four weeks following the infusion.
  Participants will record the number of hours of school attendance where relevant (e.g. no school holidays, no medical appointments).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Isaac, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No